CLINICAL TRIAL: NCT03022123
Title: The Study of Pegylated Liposomal Doxorubicin Contrast Epirubicin for the Initial Treatment of Patients With Diffuse Large B-cell Lymphoma
Brief Title: The Study of Pegylated Liposomal Doxorubicin Contrast Epirubicin for the Treatment of Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS- DLBCL -02
Record Dates: First submitted 2017-01-09; First posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-10

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Epirubicin; Prednisone; Vincristine; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pegylated liposomal doxorubicin (Experimental): PL-doxorubicin 35-40 mg/m(2) was given on day 1 in combination with standard dosage of prednisone, vincristine, cyclophosphamide (according to CHOP regimen) every 21 days for six courses;Rituximab 375 mg/m(2) was given on day 0.
  Interventions: Drug: PL-doxorubicin and epirubicin
- Epirubicin (Active Comparator): Epirubicin 70 mg/m(2) was given on day 1 in combination with standard dosage of prednisone, vincristine, cyclophosphamide (according to CHOP regimen) every 21 days for six courses;Rituximab 375 mg/m(2) was given on day 0.
  Interventions: Drug: PL-doxorubicin and epirubicin

INTERVENTIONS:
Drug: PL-doxorubicin and epirubicin — PL-doxorubicin 35-40 mg/m(2) and epirubicin 70 mg/m(2) were given in combination with standard dosage of prednisone, vincristine, cyclophosphamide, rituximab (according to CHOP-R regimen) every 21 days for six courses.
  Other Names: prednisone; vincristine; cyclophosphamide; rituximab

SUMMARY:
270 untreated patients, age between 18 and 65 years , with diffuse large B-cell lymphoma (B-DLCL) were treated with a pegylated liposomal doxorubicin (PL-doxorubicin) modiﬁed CHOP-rituximab regimen. PL-doxorubicin 35-40 mg/m(2)and epirubicin 70mg/m(2) were given in combination with standard dosage of prednisone, vincristine, cyclophosphamide, rituximab (according to CHOP-R regimen) every 21 days for six courses.

DETAILED DESCRIPTION:
PL-doxorubicin 35-40 mg/m(2) and epirubicin 70mg/m(2) were given on day 1 in combination with standard dosage of prednisone, vincristine, cyclophosphamide (according to CHOP regimen) every 21days for six courses. The choice to adopt the dosage of 30 mg/m2(instead of 50 mg/m2 of conventionaldoxorubicin) was based on pharmacokinetic data and on the results of previous studies in lymphoma.Rituximab 375 mg/m2 was given on day 0 in subsequent courses of therapy. Granulocyte colony-stimulating factor was given in the presence of grade 4 neutropenia or febrile neutropenia until hematological recovery. Treatment was stopped if lymphoma progressed, the patient refused further participation,or if there was any other intercurrent clinical condition or adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Diagnosis of previously-untreated DLBCL(patients with a transformed untreated low-grade lymphoproliferative disease were accepted)
* ECOG performance status < 3 (and higher if due to lym-phoma)
* No symptomatic cardiac arrythmias or heart failure
* Acceptable renal, hepatic and pulmonary function
* Standard laboratory and radiological staging procedures and left ventricular ejection fraction analysis by echocardiography or scintigraphy were required before therapy in all cases
* The protocol was approved by the ethics review committee of each partici- pating center
* All patients gave informed written consent.

Exclusion Criteria:

* Patients with a previous history of cardiac disease;
* HIV-HBsAg-HCV positivity, central nervous system involvement or any other major clinicalcondition;
* Other than lymphoma, which might have precluded a regular therapeutic course, were excluded from the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
overall response rate | up to 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Liu Lihong, archiater, Principal Investigator — Hebei Medical University Fourth Hospital; Liu Lihong, archiater, Study Director — Hebei Medical University Fourth Hospital
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No